CLINICAL TRIAL: NCT01818622
Title: Virtual Darkness as Additive Treatment in Mania- a Randomized Controlled Trial
Brief Title: Virtual Darkness as Additive Treatment in Mania
Acronym: VATMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Fonna (Other)
Collaborators: University of Bergen (Other); Helse Vest (Other); Moodnet (Unknown)
Responsible Party: Principal Investigator, Tone Elise Gjoetterud Henriksen, Chief Consultant, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 911678; 2011/1668 (Other: Regional Ethics Committee North)
Record Dates: First submitted 2013-03-22; First posted 2013-03-26 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar Disorder; Mania
Keywords: Bipolar disorder; Mania; Blue-blockers; Virtual darkness therapy; Actigraphy; Randomized controlled trial
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Early Detection of Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patient-group blue-blockers (Experimental): N= 21 Blue-blocking goggles/screens from 6 p.m. to 08 a.m. in addition to treatment as usual (TAU). The goggles may be taken of when going to bed and turning of the light. For consenting patients who are unable to use goggles according to the protocol blue-blocking screens covering light-sources will be used.
  Interventions: Device: Blue-blocking goggles/screens
- Patient group clear-lensed goggles (Placebo Comparator): N= 21 (Patient group) clear-lensed goggles from 06 p.m. to 08 a.m. in addition to TAU.
  Interventions: Device: Clear-lensed goggles
- Non-bipolar control-group blue-blockers (Experimental): N= 42 For baseline day 1-7: Actiwatch Spectrum worn at the wrist of dominant hand, day 8-14 continued wearing of Actiwatch spectrum + blue-blocking goggles from 6 p.m. to 08 a.m. In addition to selfreport forms described in the outcome section self report forms Horne-Ostberg Morningness-Eveningness Questionaire (HOMEQ)and Seasonal Pattern Assessment Questionaire (SPAQ).
  Interventions: Device: Blue-blocking goggles/screens

INTERVENTIONS:
Device: Blue-blocking goggles/screens — Goggles with amber tinted lenses, all model's transmittance spectra are identical. Goggles and screens are tested at Department of Physics and Technology, University of Bergen. Patients and non-bipolar controls choose model for best comfort.
  Other Names: Goggles from LowBlueLights.com, several different designs; Screens from Ganta Trading 047 Orange-red
  Arms: Non-bipolar control-group blue-blockers; Patient-group blue-blockers
Device: Clear-lensed goggles — Clear lensed safety eyewear. Patients may choose model for best comfort.
  Other Names: Uvex Genesis; Cocraft Safety Glasses 40-7362; 3M Refine 300 PC AS/AF
  Arms: Patient group clear-lensed goggles

SUMMARY:
In this randomized controlled study we will investigate the effect of blue-blocking goggles or screens (virtual darkness therapy) on manic symptoms in bipolar disorder compared to placebo. This 3-armed study includes 2 patient-groups and a non-bipolar control-group. The main hypothesis is that virtual darkness therapy is effective as additive treatment in mania.Other hypotheses are that virtual darkness therapy has significant effects on sleep, motor activity, circadian rhythm and mood also in the non-bipolar control-group.

DETAILED DESCRIPTION:
Recent discoveries in neurophysiology has shown that "virtual darkness" is achievable by blocking blue wavelengths of light (Phelps, 2007). A newly discovered retinal photoreceptor called the Intrinsically photoresponsive retinal ganglion-cell (IpRGC) whose fibers directly synapses with the suprachiasmatic nucleus (SCN), responds only to a narrow band of wavelengths with highest sensitivity between 446 and 484 nm (Brainard et al., 2001; Berson 2007). Amber tinted goggles preserve normal nocturnal melatonin levels in light environments, which means that blocking of the blue wavelengths is perceived as virtual darkness to the SCN (Kayumov, 2005; Sasseville, 2006).

In this randomized controlled study we will investigate the effect of blue-blocking goggles or screens (virtual darkness therapy) on manic symptoms in bipolar disorder compared to placebo. The general feasibility of the method both in research and treatment will be evaluated. This is a multi-site study covering Helse Fonna Local Health Authority's catchment area wich serves a population of 120000 adults. This 3-armed study includes 2 patient-groups and a non-bipolar control-group. The main hypothesis is that virtual darkness therapy is effective as additive treatment in mania.Other hypotheses are that virtual darkness therapy has significant effects on sleep, motor activity, circadian rhythm and mood also in the non-bipolar control-group. The study may contribute to develop a supplement to the current treatment in mania and may also generate new hypotheses about the underlying pathophysiological mechanisms in bipolar disorder.

ELIGIBILITY:
PATIENT GROUPS

Inclusion Criteria:

* Inpatients
* Diagnosis of DSM IV-TR of Bipolar I or Bipolar II disorder with current manic episode as verified by the semistructured interview MINI plus
* Ability to comply with the protocol
* Willingness to participate in the study
* Delayed written informed consent at discharge

Exclusion Criteria:

* Inability to comply with the protocol
* Severe retinal damage, cataract or corneal damage on both eyes
* Daily use of NSAIDS
* Daily use of betablockers
* Daily use of calcium-antagonists

NON-BIPOLAR CONTROLS

Inclusion Criteria:

* Written informed consent

Exclusion Criteria:

* Working night shift
* Diagnosed with bipolar disorder or single manic episode
* Severe retinal damage, cataract or corneal damage on both eyes
* Daily use of alcohol
* Daily use of benzodiazepines
* Daily use of NSAIDS
* Daily use of betablockers
* Daily use of calcium-antagonists

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) score | Change from baseline in YMRS score after 7 days
  The YMRS-score is assessed daily at 12 a.m. for 7 days

SECONDARY OUTCOMES:
Change in motor activity measured by use of actigraphy, Actiwatch Spectrum device | Change in motor activity over 7 days ( patients) or 14 days ( non-bipolar controls) .
  Patient-groups wear Actiwatch Spectrum for 7 days. Non-bipolar controls wear Actiwatch Spectrum for 14 days (day 1-7 for baseline, day 8-14 with intervention)

OTHER OUTCOMES:
For the non-bipolar control-group: self report forms Mood Visual Analog Scale, Positive And Negative Affect Schedule and Sleep Diary | 14 days
Self-report form for patient's experience. | At discharge
  Self report form developed for the trial for patients experience with the intervention, wearing of Actiwatch Spectrum and general participation in the trial, and section for other comments.
Self report form for non-bipolar controls on experience with intervention | At end of intervention, day 14
  3 questions: 1)Did you notice any change during the intervention? 2)If yes in question 1)When did you first notice any change? 3)If yes in question 1)Describe the experience in own words

CONTACTS AND LOCATIONS:
Overall Officials: Anders Lund, PhD, Study Director — University of Bergen, Moodnet
Locations (2):
- Norway (2):
  - Haugesund Hospital and Haugaland District Psychiatric Hospital, Haugesund
  - Valen Hospital and Folgfonn District Hospital, Valen

REFERENCES:
- [Background] Phelps J. Dark therapy for bipolar disorder using amber lenses for blue light blockade. Med Hypotheses. 2008;70(2):224-9. doi: 10.1016/j.mehy.2007.05.026. Epub 2007 Jul 16. PMID 17637502
- [Background] Berson DM. Phototransduction in ganglion-cell photoreceptors. Pflugers Arch. 2007 Aug;454(5):849-55. doi: 10.1007/s00424-007-0242-2. Epub 2007 Mar 10. PMID 17351786
- [Background] Brainard GC, Hanifin JP, Greeson JM, Byrne B, Glickman G, Gerner E, Rollag MD. Action spectrum for melatonin regulation in humans: evidence for a novel circadian photoreceptor. J Neurosci. 2001 Aug 15;21(16):6405-12. doi: 10.1523/JNEUROSCI.21-16-06405.2001. PMID 11487664
- [Background] Kayumov L, Casper RF, Hawa RJ, Perelman B, Chung SA, Sokalsky S, Shapiro CM. Blocking low-wavelength light prevents nocturnal melatonin suppression with no adverse effect on performance during simulated shift work. J Clin Endocrinol Metab. 2005 May;90(5):2755-61. doi: 10.1210/jc.2004-2062. Epub 2005 Feb 15. PMID 15713707
- [Background] Sasseville A, Paquet N, Sevigny J, Hebert M. Blue blocker glasses impede the capacity of bright light to suppress melatonin production. J Pineal Res. 2006 Aug;41(1):73-8. doi: 10.1111/j.1600-079X.2006.00332.x. PMID 16842544